CLINICAL TRIAL: NCT02782247
Title: Changes in Dynamic Liver Function Tests in Patients With Chronic Viral Hepatitis Undergoing Antiviral Therapy
Brief Title: Dynamic Liver Tests in Liver Disease
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: LAPresearch UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: 011006
Record Dates: First submitted 2016-05-06; First posted 2016-05-25 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis B; Hepatitis C
MeSH Terms: conditions — Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Short term Hepatitis C patients: 60 patients with chronic hepatitis C infection and cirrhosis who are planning to start antiviral therapy will be enrolled. Patients will be tested within 3 months prior to starting treatment. This will be repeated at 16 weeks (+/- 1 week) and again 1 calendar year after treatment initiation. Patients will have transient elastography and Indocyanine green excretion tests at each appointment.
  Interventions: Device: Transient elastography; Device: Indocyanine Green excretion
- Medium term Hepatitis C patients: 60 patients with chronic hepatitis C infection and cirrhosis who have been successfully treated in the past 3 or 5 years (+/- 3 months). Patients will have transient elastography and Indocyanine green excretion tests at each appointment.
  Interventions: Device: Transient elastography; Device: Indocyanine Green excretion
- Hepatitis B Patients: 60 patients with chronic hepatitis B and cirrhosis will be tested within 3 months prior to starting treatment. This will be repeated at 16 weeks (+/- 1 week) and again 1 calendar year after treatment initiation. Patients who have started treatment past 3 or 5 years (+/- 3 months) will also be tested. Patients will have transient elastography and Indocyanine green excretion tests at each appointment.
  Interventions: Device: Transient elastography; Device: Indocyanine Green excretion

INTERVENTIONS:
Device: Transient elastography — Transient elastography will be measured using a Fibroscan® machine which is manufactured by echosens®. It has a CE mark of 0459.
  It is a non-invasive method to accurately measure stiffness of a patient's liver without the need for a liver biopsy. This is measured by an externally placed ultrasound probe which creates an elastic shear wave at 50Hz, and measures the velocity of the echo through the liver tissue. The liver stiffness is measured in kilopascals (kPa). It has been shown to be 99% effective in detecting cirrhosis in hepatitis C and has been shown to correlate with hepatoma production in both hepatitis C and hepatitis B. Values range from - normal < 9.6 kPa, significant fibrosis 9.6-11.4kPa, cirrhosis >11.5kPa. It cannot be used in patients with ascites.
  Other Names: Fibroscan
Device: Indocyanine Green excretion — The machine to monitor the elimination of Indocyanine green is manufactured by PULSION medical systems (Munich, Germany) and consists of the PulsioFlex monitor and LiMON module. The LiMON module is a finger probe which measure near-infrared wavelengths between 805nm and 905nm. The absorption maximum for Indocyanine green is 800nm and emission at 830nm. This is then used to produce two calculations. The first is plasma disappearance rate of indocyanine green (PDRICG). This is based on working out the constant and backward extrapolation and expressed as a percentage per minute. The other is the retention ratio after 15 minutes (ICG15).
  Other Names: Pulsion Limon system

SUMMARY:
Chronic viral hepatitis often leads to liver scarring - cirrhosis. If the virus is eradicated from the liver, the liver scarring and liver function often recovers. In some patients the damage is too severe and recovery does not take place. It is not yet known which patients have liver disease that is too advanced to benefit from therapy nor is it known how fast the recovery occurs.

Non-intrusive dynamic liver testing (DLT) may allow us to predict the functionality of the liver post treatment and may guide us in treatment choices - for example patients who are predicted not to recover may be prioritised for transplantation. Indocyanine green (ICG) is a dye solely excreted by the liver into bile and used to measure its dynamic function. Transient elastography is similar to ultrasound and measures the degree of fibrosis within the liver.

The investigators hypothesise that the use of non-intrusive dynamic liver testing pre-treatment, will allow us to delineate patients before therapy who will have functional liver recovery following viral eradication.

The investigators hypothesise that monitoring changes in liver fibrosis and liver function in patients with historical viral clearance will allow an assessment of the likely speed of recovery of liver fibrosis and function - for example if all patients 5 years after treatment for viral hepatitis induced cirrhosis have 'normal' fibrosis and liver function scores the investigators will be able to conclude that recovery is complete within 5 years.

The investigators will perform a study pre and post-treatment assessing liver function using non-intrusive dynamic liver testing in addition to currently-used 'liver function' scoring systems, in a multivariate analysis, to determine whether or not the investigators can identify patients who are will have functional liver recovery post therapy.

DETAILED DESCRIPTION:
Multiple diseases affect the liver's performance, including hepatitis' B and C viruses. Hepatitis infects the liver; ultimately leading to cirrhosis associated with complications (e.g. bleeding and death), termed decompensated cirrhosis. Hepatitis induced decompensated liver disease is likely to improve upon eradication of the virus as will liver function.

Recently, Hepatitis C has seen new, more efficacious therapies, allowing functional outcomes to be evaluated following viral clearance. It has been shown this treatment regime is effective in eliminating the virus in 70% of patients but functional improvement to be 40% with the rest stagnating or becoming worse. These patients may have benefited from liver transplantation initially, followed by viral eradication therapy.

Treatment of the Hepatitis B virus is to stop more copies to be produced within cells. This on the most part is successful and the liver recovers. However, after 5 years of treatment 26% of people do not recover sufficiently and the ability to identify these early is important to their future management.

Non-intrusive dynamic liver testing (DLT) may allow us to predict the functionality of the liver post treatment and may guide us in adequate management strategies. Indocyanine green (ICG) is a dye solely excreted by the liver into bile and used to measure its dynamic function. Transient elastography is similar to ultrasound and measures the degree of fibrosis within the liver.

The investigators hypothesise the use of non-intrusive dynamic liver testing pre-treatment, will allow us to delineate patients early, who would benefit from the most intensive treatments (e.g. transplant), and spare those with less severe disease the risks and potential side effects.

The investigators will perform a study pre and post-treatment for DLT. These will be amalgamated with currently-used scoring systems, in a multivariate analysis, to ascertain the values and thus best-treatment option for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending The Royal London Hospital with cirrhosis (defined as fibroscan score >11.5 OR aspartate aminotransferase (AST) to platelet ratio index (APRI) score >2 OR liver biopsy or imaging report of cirrhosis) who are planning to commence antiviral therapy for either chronic hepatitis B or chronic hepatitis C.
* Patients attending The Royal London Hospital with cirrhosis (defined as above) due to chronic hepatitis C infection who have undergone successful antiviral therapy in the past.
* Patients attending The Royal London Hospital with cirrhosis (defined as above) due to chronic hepatitis B infection who are taking antiviral medication
* Age 18 or above
* Willing and able to provide Informed consent

Exclusion Criteria:

* Any inclusion criteria not met
* Pregnancy or breast feeding
* Known allergy to ICG

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential patients will be seen in clinic by their clinical team and will come to an agreement with regard to the treatment options available to them. Those that meet the above criteria will then be offered the opportunity to partake in research with the understanding these tests will not affect their treatment in any way. They will be referred to the research team for informed consent to be taken.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline following 1 year of treatment for chronic viral hepatitis with cirrhosis using transient elastography. | Baseline, 4 months and 1 year
  Patients are treated for hepatitis B or hepatitis C and tested at baseline, 4 months and 1 year. Scores range from 0 to 75kPa with cirrhosis defined as above 11.5kPa. Change in baseline is noted. (Change = 4 month or 1 year measurement - baseline).
Change from baseline following 1 year of treatment for chronic viral hepatitis with cirrhosis using indocyanine green excretion test using plasma disappearance rate. | Baseline, 4 months and 1 year
  Patients are treated for hepatitis B or hepatitis C and tested at baseline, 4 months and 1 year. Measurement of plasma disappearance rate of Indocyanine green (PDRicg) is measured with normal between 18-25%/min. Change in baseline is noted.
Change from baseline following 1 year of treatment for chronic viral hepatitis with cirrhosis using indocyanine green excretion test using plasma retention rate at 15 minutes. | Baseline, 4 months and 1 year
  Patients are treated for hepatitis B or hepatitis C and tested at baseline, 4 months and 1 year. Measurement of retention rate of indocyanine green at 15 minutes is measured (ICG15) with normal being below 10%. Change in baseline is noted.

SECONDARY OUTCOMES:
Percentage of participants achieving normal fibroscan and or indocyanine green excretion test results at 3 or 5 years post initiation of treatment for viral hepatitis. | 3 years, 5 years
  Patients treated for hepatitis B or hepatitis C with cirrhosis are tested at either 3 or 5 years after initiation of treatment. Fibroscan, score (range from 0 to 75kPa with cirrhosis defined as above 11.5kPa), measurement of plasma disappearance rate of Indocyanine green (PDRicg) (normal between 18-25%/min) and measurement of retention rate of indocyanine green at 15 minutes is measured (ICG15) (normal below 10%) are tested with the percentage of patients achieving normal in all tests reported.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Foster, PhD, MBBS, Principal Investigator — Queen Mary University of London
Locations (1):
- Bart's Health NHS, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marcellin P, Gane E, Buti M, Afdhal N, Sievert W, Jacobson IM, Washington MK, Germanidis G, Flaherty JF, Aguilar Schall R, Bornstein JD, Kitrinos KM, Subramanian GM, McHutchison JG, Heathcote EJ. Regression of cirrhosis during treatment with tenofovir disoproxil fumarate for chronic hepatitis B: a 5-year open-label follow-up study. Lancet. 2013 Feb 9;381(9865):468-75. doi: 10.1016/S0140-6736(12)61425-1. Epub 2012 Dec 10. PMID 23234725
- [Background] Gupta S, Chawla Y, Kaur J, Saxena R, Duseja A, Dhiman RK, Choudhary NS. Indocyanine green clearance test (using spectrophotometry) and its correlation with model for end stage liver disease (MELD) score in Indian patients with cirrhosis of liver. Trop Gastroenterol. 2012 Apr-Jun;33(2):129-34. doi: 10.7869/tg.2012.30. PMID 23025060
- [Background] Wilder J, Patel K. The clinical utility of FibroScan((R)) as a noninvasive diagnostic test for liver disease. Med Devices (Auckl). 2014 May 3;7:107-14. doi: 10.2147/MDER.S46943. eCollection 2014. PMID 24833926
- [Background] Faybik P, Hetz H. Plasma disappearance rate of indocyanine green in liver dysfunction. Transplant Proc. 2006 Apr;38(3):801-2. doi: 10.1016/j.transproceed.2006.01.049. PMID 16647475
- [Background] Procopet B, Berzigotti A, Abraldes JG, Turon F, Hernandez-Gea V, Garcia-Pagan JC, Bosch J. Real-time shear-wave elastography: applicability, reliability and accuracy for clinically significant portal hypertension. J Hepatol. 2015 May;62(5):1068-75. doi: 10.1016/j.jhep.2014.12.007. Epub 2014 Dec 13. PMID 25514554
- [Background] Foster GR, Irving WL, Cheung MC, Walker AJ, Hudson BE, Verma S, McLauchlan J, Mutimer DJ, Brown A, Gelson WT, MacDonald DC, Agarwal K; HCV Research, UK. Impact of direct acting antiviral therapy in patients with chronic hepatitis C and decompensated cirrhosis. J Hepatol. 2016 Jun;64(6):1224-31. doi: 10.1016/j.jhep.2016.01.029. Epub 2016 Jan 30. PMID 26829205